CLINICAL TRIAL: NCT03746769
Title: Improving Islet Transplantation Outcomes With Gastrin
Brief Title: Improving Islet Transplantation Outcomes With Gastrin for Type I Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18156
Record Dates: First submitted 2018-11-09; First posted 2018-11-20 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: islet; islet cell; transplant; gastrin; hypoglycemia; labile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — gastrin 17

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental)
  Interventions: Biological: Allogenic Human Islet Cells; Drug: Gastrin 17

INTERVENTIONS:
Biological: Allogenic Human Islet Cells — islet cells transplanted into the portal vein in the liver
Drug: Gastrin 17 — Gastrin-17 (or GAST-17) - a gut hormone injected under the skin twice daily for 30 days soon after islet transplant and again 6 months later.
  Also, anti-rejection medications (to prevent the body from rejecting the islet cells) and other medications to guard against infection and support participant health and/or the health of the transplanted islets.

SUMMARY:
This clinical study will evaluate the safety and effectiveness of Gastrin treatment with islet transplantation to help patients with difficult to control type 1 diabetes make insulin again and improve blood sugar control.

This study involves two investigational (experimental) products not yet approved by the U.S. Food and Drug Administration (FDA) as a treatment for any disease:

1. Human allogenic islet cells (islet cells from a deceased, unrelated human donor)
2. Gastrin-17 (Gastrin) - a hormone secreted by the gut

DETAILED DESCRIPTION:
Islet cell transplantation involves transplanting the cells that make insulin from a pancreas of deceased organ donor to a patient with diabetes. Because there is a limited supply of donor islet cells available, this study is testing whether Gastrin injections can help make a fewer number of transplanted islets work better.

Gastrin is a natural gut hormone that is present in the pancreas during its development in the embryo but not after birth, and is believed to participate in the formation of the normal pancreas. Several studies have tried to use gastrin to help grow insulin making islet cells in laboratory experiments or after transplanting islets in laboratory animals. In early clinical trials, diabetic patients treated with gastrin and other growth factors required less insulin after 4 weeks of gastrin treatment and the effect lasted more than 12 weeks after stopping treatment, suggesting that gastrin may have increased the number of cells that make insulin.

This study will evaluate whether taking Gastrin injections following a single islet transplantation is safe, improves how well the islet transplant works and/or helps increase the number of insulin-making cells in the islets.

Qualified participants will receive treatment with a single islet transplant and two rounds of gastrin treatment (twice daily injections for 30 days) with transplant and again 6 months later. Study participants will also take anti-rejection medications (to prevent the body from rejecting the islet cells) and other medications to guard against infection and support their health and/or the health of the transplanted islets. Participants will need to return to City of Hope in Duarte, CA for frequent follow-up visits for one year after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-68 years
2. Type 1 diabetes mellitus (documented with fasting C-peptide level of </= 0.2 ng/ml before and </= 0.3 ng/ml after IV administration of 1 mg of glucagon) for at least 5 years.
3. Unstable blood glucose characterized by:

   Frequent hypoglycemia (blood glucose less than or equal to 54 mg/dl more than once per week)

   -and/or- Hypoglycemia unawareness (Clarke score of 4 or more).

   -and/or- One or more severe hypoglycemic episodes in 12 months preceding enrollment

   -and/or- Erratic blood glucose levels that interfere with daily activities

   -and/or- One or more hospital visits for diabetic ketoacidosis in the 12 months preceding enrollment
4. Ability and willingness to comply with post-transplant regimen, including immunosuppression, use of reliable contraception, frequent clinic visits, testing and maintaining detailed logs of blood glucose levels, insulin doses and medications, and completing detailed follow-up studies.
5. Ability to give informed consent.
6. Fully vaccinated against COVID-19

Exclusion Criteria:

1. BMI > 33
2. Insulin requirements > 1.0 units/kg/day
3. Significant kidney disease (estimated GFR from serum creatinine measurement <65 ml/min, random spot urine microalbumin to creatinine ratio >300mg albumin/g creatinine)
4. Significant hepatobiliary disease, including elevation of liver enzymes > twice the upper limit of normal for each of ALT and AST (any elevation of these enzymes will be determined), bilirubin not within normal limits, albumin < 3.5 g/dl, liver masses, portal vein thrombosis, evidence of portal hypertension, or significant, untreated gallbladder disease (i.e. gallstones)
5. Significant cardiovascular disease, including non-correctable coronary artery disease with ejection fraction < 50% and/or recent myocardial infarction (within last 12 months); or extensive peripheral vascular disease not correctable by surgery,
6. Evidence of active proliferative retinopathy
7. Hypertension( >/= 140/90) despite appropriate treatment
8. Hyperlipidemia (total cholesterol > 260 mg/dl, LDL > 160 mg/dl, and/or triglycerides > 300 mg/dl) despite appropriate treatment
9. Anemia (Hgb < 11 g/dl) or other hematologic disorders that require medical attention
10. WBC <3,000/ul
11. Increased risk of bleeding (platelet count < 120,000 cells/ul; INR > 1.5), other chronic hemostasis disorders, or treatment with chronic anticoagulant therapy (i.e. heparin or warfarin)
12. Recent unresolved acute infection (except for mild skin infection or nail fungal infection), or chronic infection, including tuberculosis, HIV, HBV, HCV, CMV or syphilis (RPR)
13. EBV IgG negative
14. Any history of malignancy, except completely resected squamous or basal cell skin cancer or in situ cancer of the cervix
15. Evidence of active peptic ulcer disease
16. History of gastric bypass
17. Recent history of non-adherence to recommended medical therapy
18. Psychiatric illness that is untreated, or likely to interfere significantly with study compliance despite treatment
19. Previous organ/tissue transplant
20. Administration of live attenuated vaccines within 60 days of enrollment.
21. Presence of a chronic disease that must be chronically treated with contraindicated medications
22. Use of investigational agents within four weeks of enrollment
23. Active alcohol or substance abuse, including cigarette smoking (must be abstinent for > 3 months)
24. Pregnant women, women intending future pregnancy, women of reproductive potential who are unable or unwilling to follow effective contraceptive measures (i.e., tubal ligation, two barrier methods, abstinence) for the duration of study treatment and for as long as they are on immunosuppressive medication, and women presently breastfeeding.
25. Individuals without health insurance covering the cost of immunosuppression and clinical and laboratory follow-up after completion of the study
26. Any medical condition that in the opinion of the investigator will interfere with safe participation in the trial

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-07 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who are insulin independent, free from severe hypoglycemia and have HbA1c less than or equal to 6.5% ("complete response") | 1 year post transplant (6 months after second course of Gastrin)

SECONDARY OUTCOMES:
Proportion of subjects who are free of severe hypoglycemic episodes (SHE) and have a HbA1c less than or equal to 7.0% ("partial response"). | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course

OTHER OUTCOMES:
Reduction/elimination of hypoglycemia | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Reduction in daily insulin use | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Reduction of daily insulin use per 100,000 IEQ transplanted | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
C-peptide/insulin secretion response to glucose/arginine stimulation and other metabolic studies. | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Incidence of treatment-related adverse events | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Incidence of a change in immunosuppression drug regimen | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
The incidence of immune sensitization defined by presence of anti-HLA antibodies absent prior to transplant | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Incidence of discontinuation of immunosuppression | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Incidence of change or early discontinuation of Gastrin treatment | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Incidence of change or early discontinuation of sitagliptin/esomeprazole supportive therapy | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Improvement in glucose time in range during continuous glucose monitoring | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course
Improvement in Personal Glycemic State (PGS) score calculated from continuous glucose monitoring | At Month 1, Month 2.5, and Month 6 post start of each Gastrin course

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- See also: City of Hope Islet Cell Transplantation Program — https://www.cityofhope.org/islets